CLINICAL TRIAL: NCT02929810
Title: Lowering Blood Pressure by Sleep Extension: a Randomized, Controlled Trial
Brief Title: Sleep Extension and Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Virend Somers, MD, PhD, Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-000987
Record Dates: First submitted 2016-10-09; First posted 2016-10-11 (Estimated); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Sleep Extension

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sleep extension (Experimental)
  Interventions: Behavioral: sleep extension
- sleep maintenance (Active Comparator)
  Interventions: Behavioral: sleep maintenance

INTERVENTIONS:
Behavioral: sleep extension
  Arms: sleep extension
Behavioral: sleep maintenance
  Arms: sleep maintenance

SUMMARY:
Emerging evidence suggests that approximately 30% of the US adult population sleeps less than 7 hours per night, and those who do exhibit 20-52% enhanced risk to develop cardiovascular diseases and particularly hypertension. Since sleep curtailment is largely voluntary, sleep deficiency can be corrected and its detrimental health consequences potentially reversed. The purpose of the present proposal is to investigate the cardiovascular and metabolic effects of sleep extension in prehypertensive and stage 1 hypertensive subjects who report habitual short sleep.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 65 (inclusive)
* Gender: both males and females
* Body mass index (BMI): 18.5-34.9 kg/m2
* Habitual sleep duration: <7 hours
* Presence of either:

  * Prehypertension: office systolic BP (SBP) 120-139 mmHg and/or diastolic BP (DBP) 80- 89 mmHg;
  * Stage 1 hypertension: office SBP 140-159 mmHg and/or DBP 90-99 mmHg
* Either on no prescription medications (other than oral contraceptive pills, or intrauterine devices) or on stable medical regimen for at least 1 month, if taking prescription medications for chronic conditions
* Not pregnant or breast feeding and not intending to become pregnant or breast feed
* Not a current smoker or tobacco user
* Ability to provide written informed consent

Exclusion Criteria:

* Vulnerable study populations will be excluded
* Pregnancy
* Smoking
* Presence of overt cardiovascular diseases, diabetes, chronic kidney disease, cancer, sleep disorders, psychiatric disorders
* If taking prescription medications for chronic conditions, change in therapy (type, frequency and/or dosage) over the previous month
* Habitual sleep duration ≥7 hours
* Excessive alcohol (≥15 drinks/week in men and ≥8 drinks/week in women) and/or excessive caffeine intake (>400 mg)
* Currently on a diet and/or actively trying to lose weight
* Currently or previously (during the past 2 months) participation in any other research study at the discretion of study personnel
* Blood/plasma donation during the past 2 months
* Unwillingness or inability to adjust sleep schedule.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-10; Primary Completion 2023-09-07 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
change in 24-hour mean arterial pressure | 8 weeks

SECONDARY OUTCOMES:
change in baroreflex sensitivity | 8 weeks
change in endothelial function | 8 weeks
change in insulin sensitivity | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Virend Somers, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials